CLINICAL TRIAL: NCT01653171
Title: Effectiveness of Premedication With Simethicone or Simethicone Plus N-acetylcysteine vs. Placebo in Improving Visibility During Upper Endoscopy.
Brief Title: Premedication With Simethicone or Simethicone Plus N-acetylcysteine in Improving Visibility During Upper Endoscopy
Acronym: PRUE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Hugo Monrroy, Internal Medicine Physician, Gastroenterology Residency Training Program, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 12-221
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Stomach Neoplasms
Keywords: Acetylcysteine, Simethicone, Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Water; Simethicone; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Control (No Intervention): Standard upper endoscopy withouth premedication
- Water (Placebo Comparator): 100 mL of water, 20 minutes before upper endoscopy
  Interventions: Drug: Water (Placebo)
- Simethicone (Experimental): Simethicone 200 mg, in water for up to 100 mL, to take 20 minutes prior to examination
  Interventions: Drug: Simethicone
- N-acetylcysteine 500 mg + Simethicone (Experimental): N-acetylcysteine 500 mg + Simethicone 200 mg in water for up to 100 mL, to take 20 minutes prior to examination
  Interventions: Drug: Simethicone; Drug: N-acetylcysteine 500 mg
- N-acetylcysteine 1000 mg + Simethicone (Experimental): N-acetylcysteine 1000 mg + Simethicone 200 mg in water for up to 100 mL, to take 20 minutes prior to examination
  Interventions: Drug: Simethicone; Drug: N-acetylcysteine 1000 mg

INTERVENTIONS:
Drug: Water (Placebo) — Water 100 mL
  Other Names: (Placebo)
  Arms: Water
Drug: Simethicone — 200 mg (5 mL) in water for up to 100 mL, to take 20 minutes prior to examination
  Other Names: Flapex, Andromaco, Chile
  Arms: N-acetylcysteine 1000 mg + Simethicone; N-acetylcysteine 500 mg + Simethicone; Simethicone
Drug: N-acetylcysteine 500 mg — 500 mg + Simethicone 200 mg in water for up to 100 mL, to take 20 minutes prior to examination
  Other Names: Mucolítico, Sanitas, Chile
  Arms: N-acetylcysteine 500 mg + Simethicone
Drug: N-acetylcysteine 1000 mg — 1000 mg + Simethicone 200 mg in water for up to 100 mL, to take 20 minutes prior to examination
  Other Names: Mucolítico, Sanitas, Chile
  Arms: N-acetylcysteine 1000 mg + Simethicone

SUMMARY:
The purpose of this study is to determine whether premedication with Simethicone or Simethicone plus N-acetylcysteine are effective improving visibility during Upper endoscopy compared with use of water or no preparation.

DETAILED DESCRIPTION:
While globally there has been a downward trend in the incidence of gastric cancer, it remains the second leading cause of cancer mortality in the world. In Chile is the leading cause of death from malignant tumors in both sexes, and is recognized as a problem and public health priority in our country. Detection of gastric cancer in early stages has a huge impact on healing and therefore the prognosis of patients. In countries like Japan, where the incidence of this neoplasm is one of the highest in the world, mass screening programs have failed to demonstrate significant impact at the population level, there is a body of evidence to support endoscopic screening especially with the advent of new minimally invasive procedures such as endoscopic mucosal resection for gastric cancers detected in early stages. In our country, it is estimated that about half of the patients already have lymph node metastases or involvement of adjacent organs at diagnosis. The best way to reduce disease burden from this disease would be through primary prevention interventions or effective early detection. For this purpose the upper gastrointestinal endoscopy is the method of choice to examine the gastric mucosa in search of early lesions, and this is the point where adequate visibility of the mucosa is overriding. Mucus, foam and bubbles accumulated in the gastrointestinal tract mucosa interfere with adequate endoscopic visualization and thus represent risk of failing to diagnose early lesions. For this reason is that various anti-foam agents, anti-bubbles are widely used in endoscopic centers mainly in Japan, where its use is almost a rule, unlike the West where its use is limited by the theoretical risk of aspiration. Simethicone has been proven as a good anti-foam agent prior to endoscopy to remove mucus and bubbles. It has also been studied in other scenarios such as colonoscopy as an additive in the preparation of the colon to eliminate bubbles in endoscopic capsule for small bowel preparation as well as Endoscopic Ultrasound which reduces artifacts and increases the accuracy of the study. Currently N-acetylcysteine, a mucolytic agent, either alone or in combination with Simethicone has proven effective in removing mucus and gastric bubbles when used 20 minutes prior to the upper endoscopy, improving the visualization of the gastric mucosa. Other agents such as pronase have also been described as useful in this task are not yet available in our area. In the context of the relevance of gastric cancer in our environment, our low rate of early cancer detection and the absence of national policies on the preparation and agents that may improve visualization of the mucosa, this study aims to compare the effect of products available in our country in preparation for an endoscopy in order to improve visualization of the mucosa and increase the chance of recognizing early lesions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic upper endoscopy performed for medical indications

Exclusion Criteria:

* Upper gastrointestinal surgery
* Gastric Cancer
* Deep sedation with propofol
* Indication of therapeutic endoscopy
* Emergency endoscopy
* Patients with a history of

  * Upper gastrointestinal bleeding
  * Caustic ingestion
  * Pregnancy
  * Diabetes mellitus
  * Asthma
  * Allergic reactions to medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Visibility at upper endoscopy | During diagnostic upper endoscopy
  The antrum, proximal part of the greater curvature, distal part of the greater curvature and the gastric fundus were assessed separately in terms of visibility mucosa. He scored from 1 to 4 each zone according to a score of visibility, as defined in previous publications by Chang et al. The sum of the scores from the four locations was defined as the total mucosal visibility score (TMVS) for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Parra-Blanco, MD, Study Director — Pontificia Universidad Catolica de Chile; Esteban Glasinovic, MD, Principal Investigator — Pontificia Universidad Catolica; Hugo Monrroy, MD, Principal Investigator — Pontificia Universidad Catolica de Chile; Roberto Candia, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Result] Lambert R, Guilloux A, Oshima A, Pompe-Kirn V, Bray F, Parkin M, Ajiki W, Tsukuma H. Incidence and mortality from stomach cancer in Japan, Slovenia and the USA. Int J Cancer. 2002 Feb 20;97(6):811-8. doi: 10.1002/ijc.10150. PMID 11857360
- [Result] Csendes A, Smok G, Medina E, Salgado I, Rivera R, Quitral M. [Clinical course characteristics of gastric cancer 1958-1990]. Rev Med Chil. 1992 Jan;120(1):36-42. Spanish. PMID 1305308
- [Result] McColl KE. Screening for early gastric cancer. Gut. 2005 Jun;54(6):740-2. doi: 10.1136/gut.2004.058461. No abstract available. PMID 15888773
- [Result] Tashiro A, Sano M, Kinameri K, Fujita K, Takeuchi Y. Comparing mass screening techniques for gastric cancer in Japan. World J Gastroenterol. 2006 Aug 14;12(30):4873-4. doi: 10.3748/wjg.v12.i30.4873. PMID 16937471
- [Result] Everett SM, Axon AT. Early gastric cancer: disease or pseudo-disease? Lancet. 1998 May 2;351(9112):1350-2. doi: 10.1016/s0140-6736(98)04365-7. No abstract available. PMID 9643813
- [Result] Ono H, Kondo H, Gotoda T, Shirao K, Yamaguchi H, Saito D, Hosokawa K, Shimoda T, Yoshida S. Endoscopic mucosal resection for treatment of early gastric cancer. Gut. 2001 Feb;48(2):225-9. doi: 10.1136/gut.48.2.225. PMID 11156645
- [Result] Chavez Rossell M. [Endoscopic treatment of early gastric cancer: from Endoscopic Mucosal Resection (EMR) to Endoscopic Submucosal Dissection (ESD)]. Rev Gastroenterol Peru. 2005 Jan-Mar;25(1):76-92. Spanish. PMID 15818423
- [Result] Federation nationale des centres de lutte contre le cancer. [Recommendations for clinical practice: 2004 Standards, Options and Recommendations for management of patients with adenocarcinomas of the stomach (excluding cardial and other histological forms of cancer) Federation nationale des centres de lutte contre le cancer]. Gastroenterol Clin Biol. 2005 Jan;29(1):41-55. doi: 10.1016/s0399-8320(05)80692-x. No abstract available. French. PMID 15738894
- [Result] Yoon H, Kim N, Lee HS, Shin CM, Park YS, Lee DH, Park DJ, Kim HH, Jung HC. Effect of endoscopic screening at 1-year intervals on the clinicopathologic characteristics and treatment of gastric cancer in South Korea. J Gastroenterol Hepatol. 2012 May;27(5):928-34. doi: 10.1111/j.1440-1746.2011.07038.x. PMID 22142434
- [Result] Bhandari P, Green S, Hamanaka H, Nakajima T, Matsuda T, Saito Y, Oda I, Gotoda T. Use of Gascon and Pronase either as a pre-endoscopic drink or as targeted endoscopic flushes to improve visibility during gastroscopy: a prospective, randomized, controlled, blinded trial. Scand J Gastroenterol. 2010 Mar;45(3):357-61. doi: 10.3109/00365520903483643. PMID 20148732
- [Result] McDonald GB, O'Leary R, Stratton C. Pre-endoscopic use of oral simethicone. Gastrointest Endosc. 1978 Nov;24(6):283. doi: 10.1016/s0016-5107(78)73542-x. No abstract available. PMID 365670
- [Result] Banerjee B, Parker J, Waits W, Davis B. Effectiveness of preprocedure simethicone drink in improving visibility during esophagogastroduodenoscopy: a double-blind, randomized study. J Clin Gastroenterol. 1992 Oct;15(3):264-5. No abstract available. PMID 1479177
- [Result] McNally PR, Maydonovitch CL, Wong RK. The effectiveness of simethicone in improving visibility during colonoscopy: a double-blind randomized study. Gastrointest Endosc. 1988 May-Jun;34(3):255-8. doi: 10.1016/s0016-5107(88)71324-3. PMID 3292345
- [Result] Tongprasert S, Sobhonslidsuk A, Rattanasiri S. Improving quality of colonoscopy by adding simethicone to sodium phosphate bowel preparation. World J Gastroenterol. 2009 Jun 28;15(24):3032-7. doi: 10.3748/wjg.15.3032. PMID 19554657
- [Result] Albert J, Gobel CM, Lesske J, Lotterer E, Nietsch H, Fleig WE. Simethicone for small bowel preparation for capsule endoscopy: a systematic, single-blinded, controlled study. Gastrointest Endosc. 2004 Apr;59(4):487-91. doi: 10.1016/s0016-5107(04)00003-3. PMID 15044883
- [Result] Fang YH, Chen CX, Zhang BL. Effect of small bowel preparation with simethicone on capsule endoscopy. J Zhejiang Univ Sci B. 2009 Jan;10(1):46-51. doi: 10.1631/jzus.B0820148. PMID 19198022
- [Result] Chang CC, Chen SH, Lin CP, Hsieh CR, Lou HY, Suk FM, Pan S, Wu MS, Chen JN, Chen YF. Premedication with pronase or N-acetylcysteine improves visibility during gastroendoscopy: an endoscopist-blinded, prospective, randomized study. World J Gastroenterol. 2007 Jan 21;13(3):444-7. doi: 10.3748/wjg.v13.i3.444. PMID 17230616
- [Result] Kuo CH, Sheu BS, Kao AW, Wu CH, Chuang CH. A defoaming agent should be used with pronase premedication to improve visibility in upper gastrointestinal endoscopy. Endoscopy. 2002 Jul;34(7):531-4. doi: 10.1055/s-2002-33220. PMID 12170403
- [Result] Sanchez del Rio A, Alarcon Fernandez O, Baudet JS, Sainz Menendez Z, Socas Mendez M. Reliability of the Spanish version of a brief questionnaire on patient satisfaction with gastrointestinal endoscopy. Rev Esp Enferm Dig. 2005 Aug;97(8):554-61. doi: 10.4321/s1130-01082005000800003. English, Spanish. PMID 16266222
- [Result] Principles of training in gastrointestinal endoscopy. From the ASGE. American Society for Gastrointestinal Endoscopy. Gastrointest Endosc. 1999 Jun;49(6):845-53. No abstract available. PMID 10343249